CLINICAL TRIAL: NCT07242326
Title: SNAP AF-52 - An Ambidirectional Observational Study to Assess Label-Concordant Dosing and Medication Adherence (Proportion of Days Covered) for Oral Anticoagulants in Adults Aged ≥65 Years With Atrial Fibrillation Managed in Family Health Centers in Ordu, Türkiye, With Same-Day Tertiary Cardiology Referral for Unsafe Findings
Brief Title: SNAP AF-52: Dose Appropriateness and Adherence to Oral Anticoagulation in Adults ≥65 With Atrial Fibrillation in Primary Care (Ordu, Türkiye)
Acronym: SNAP AF-52
Status: Not yet recruiting | Type: Observational
Sponsor: Kotyora Family Medicine Health Management and Education Association (Network)
Collaborators: Ordu University Faculty of Medicine, Department of Cardiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: KAHSED-002; KAHSED-002 (Other: Kotyora Family Medicine Health Management and Education Association (KAHSED)); pending (Other: Ordu University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Medication Adherence; Atrial Fibrillation (AF); Direct Oral Anticoagulants (DOACs)
Keywords: DOAC;; apixaban; rivaroxaban; dabigatran; edoxaban; dose appropriateness; label-concordant dosing; Proportion of Days Covered (PDC); primary nonadherence; ISTH major bleeding; primary care
MeSH Terms: conditions — Medication Adherence; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Records Cohort: Adults aged ≥65 years with atrial fibrillation and any oral anticoagulant use documented within Dec 1, 2024-Nov 30, 2025. Data are abstracted from existing records to determine dose appropriateness at the index regimen and 12-month PDC, and to capture ischemic (I63/G45/I74) and hemorrhagic (I60-I62; ISTH major) events. No patient contact and no protocol-assigned treatment.

SUMMARY:
SNAP AF-52 is an ambidirectional observational registry conducted in family health centers (primary care) across Ordu, Türkiye, enrolling adults ≥65 years with a pre-existing diagnosis of atrial fibrillation. The study assesses (a) label-concordant dosing of oral anticoagulants (DOACs/warfarin) using drug-specific criteria, and (b) medication adherence via Proportion of Days Covered (PDC) over the prior 12 months (good adherence defined as PDC ≥80%). Unsafe findings (e.g., suspected under-/overdosing, critical drug-drug interactions, very low renal function) trigger same-day referral to tertiary cardiology for evaluation and management. The retrospective window is Dec 1, 2024-Nov 30, 2025; the prospective single-visit inclusion window is Dec 1, 2025-May 31, 2026. No experimental treatment is administered; all care is routine.

DETAILED DESCRIPTION:
Family physicians will screen their ≥65-year attendees with documented AF and record a minimum dataset during a single routine visit: demographics, body weight, most recent serum creatinine (date/value) to compute Cockcroft-Gault creatinine clearance (CrCl), current oral anticoagulant and regimen, common interacting drugs, and pharmacy dispensing dates with days' supply for the last 12 months. The system auto-classifies dose appropriateness per drug label criteria (including apixaban reduction rules; rivaroxaban/dabigatran/edoxaban CrCl thresholds and P-gp/CYP3A4 interactions) and computes PDC with carry-over of early refills; primary nonadherence is defined as no fill within 30 days of the first prescription. Retrospective capture of events includes ischemic stroke/TIA/systemic embolic event (SEE) and hemorrhagic stroke/ISTH major bleeding, plus on-treatment status at the event date.

Participants with potentially unsafe dosing or clinically high-risk interaction (e.g., strong inducers; strong dual inhibitors) or CrCl <15 mL/min are same-day referred to tertiary cardiology. Identifiable data will be stored securely per ethics approval and Turkish data protection (KVKK); only aggregated results will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years.
* Established atrial fibrillation (any type) documented in the medical record.
* Presenting to a family health center (primary care) in Ordu province during the prospective window or having records within the retrospective window.
* On an oral anticoagulant (DOAC) at any time in the 12-month window.

Exclusion Criteria:

* Mechanical prosthetic heart valve or moderate-to-severe rheumatic mitral stenosis
* Participation in an interventional drug study affecting anticoagulation
* Lack of minimal data elements required for dose classification (age, sex, body weight, serum creatinine with date, current OAC and regimen)
* Investigator judgment that reliable data cannot be obtained from records

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged ≥65 years with established atrial fibrillation (any type) receiving care in family health centers across Ordu, Türkiye. The prospective cohort enrolls consecutive eligible attendees during Dec 1, 2025-May 31, 2026 at a single routine visit; the retrospective cohort includes patients with AF who received an oral anticoagulant during Dec 15, 2025-May 31, 2026 identified from primary care records. Exclusions: mechanical prosthetic heart valve or moderate-severe rheumatic mitral stenosis, and cases lacking the minimal data needed for dose/adherence classification. No investigational treatment is delivered; care is routine with same-day tertiary referral when unsafe dosing, high-risk drug interactions, or very low renal function are detected.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1: Label-Concordant Dose Proportion | At index visit (assessed using baseline variables and the most recent renal function).
  Proportion of patients on label-concordant dose vs underdose vs overdose, by anticoagulant. Criteria include:
  Apixaban: 5 mg BID (standard) or 2.5 mg BID if ≥2 of: age ≥80 years, weight ≤60 kg, serum creatinine ≥1.5 mg/dL.
  Rivaroxaban: 20 mg QD if CrCl ≥50 mL/min; 15 mg QD if CrCl 15-49; avoid/evaluate if CrCl <15.
  Dabigatran: 150 mg BID (standard); 110 mg BID considered if age ≥80 or if CrCl 30-50 and P-gp inhibitor; avoid/evaluate if CrCl <30.
  Edoxaban: 60 mg QD (standard); 30 mg QD if CrCl 15-50, weight ≤60 kg, or specific P-gp inhibitors (e.g., dronedarone, verapamil, erythromycin, ketoconazole, cyclosporine); consider reduced efficacy if CrCl >95.
Primary Outcome 2: Good Adherence (PDC ≥80%) | Prior 12 months relative to index date
  Proportion of Days Covered (PDC) = (covered days / 365), with early refill carry-over and single-day duplicate fills not double-counted. Good adherence: PDC ≥80% (class-level and drug-specific PDC reported).

SECONDARY OUTCOMES:
Secondary Outcome 1: Primary Nonadherence | From first prescription within the 12-month
  Yes if no pharmacy dispensing within 30 days of the first OAC prescription.
Secondary Outcome 2: Ischemic Events | Prior 12 months.
  Proportion with ischemic stroke (ICD-10 I63.x), TIA (G45.x), or systemic arterial embolic event (I74.x); event-date on-treatment status derived from dispensing coverage.
Secondary Outcome 3: Hemorrhagic Events | Prior 12 months
  Hemorrhagic stroke (I60-I62) and ISTH major bleeding (any of: fatal; critical site-including intracranial/intraspinal/intraocular/pericardial/intra-articular/intramuscular with compartment syndrome; Hb drop ≥2 g/dL; or ≥2 RBC units transfused). Location examples: GI (K92.2; K25-K28 with hemorrhage), GU (R31/N02), pulmonary (R04.2), intra-ocular (H43.1/H35.6).
Secondary Outcome 4: Same-Day Tertiary Referral Rate | At index visit
  Proportion referred same-day to tertiary cardiology due to unsafe dose, high-risk interaction (e.g., strong inducer/strong dual inhibitor), or CrCl <15 mL/min.

CONTACTS AND LOCATIONS:
Overall Officials: Seçkin Dereli, MD, Assoc. Prof., Principal Investigator — Ordu University Faculty of Medicine, Department of Cardiology (Turkey)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because identifiers are retained in the working dataset to enable same-day clinical referral and safety follow-up, and the ethics approval (and patient permissions) limit use to quality-of-care evaluation within participating centers. De-identification sufficient for public sharing would require extensive linkage files and could still pose re-identification risk in a single-province cohort under local data-protection law (KVKK). We will share only aggregated, de-identified results (tables/figures) upon reasonable request and after ethics approval; the study protocol, CRF, and PDC calculation SOP can be provided as supporting documents.